CLINICAL TRIAL: NCT04932681
Title: Evaluation of the Use of Medicinal Plants and Other Alternative and Complementary Medicines by Patients With Cancer in Reunion Island
Brief Title: Use of Medicinal Plants and Other Alternative and Complementary Medicines by Patients With Cancer in Reunion Island
Acronym: CAMUCRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: APLAMEDOM (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/05
Record Dates: First submitted 2021-05-18; First posted 2021-06-21 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qualitative group: Interview about the use of Complementary and Alternative Medecine
- Quantitative group: Questionnaire about the use of Complementary and Alternative Medecine

SUMMARY:
Exploratory, observational and cross-sectional study with the aim of describing the use of plants for medicinal purposes (and other Complementary and Alternative Medicine) and identifying the determinants of this use. The methodology envisaged is mixed with an exploratory design combining qualitative (interviews) and quantitative techniques (questionnaires).

To knowledge of investigators, no study has been carried out in Reunion Island on the use of plants and other alternative and complementary medicines among cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Living in Reunion Island
* Suffering from cancer (solid tumors, hematological malignancies)
* Able to answer a questionnaire
* Patient who does not oppose to the research

Exclusion Criteria:

* Person of legal age under guardianship or under legal protection
* Persons who do not understand French or Reunionese Creole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer linving in the Reunion Island
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Use of herbal medicine | Day 1
  Proportion of patients using herbal medicine (from the patient's perspective) among cancer patients.

SECONDARY OUTCOMES:
Barriers of dialogue between patient and practionner | Day 1
  Interviews between patient and interviewer will help to extract the barriers limiting patient/practitioner dialogue on Complementary and Alternative Medicine use from patient and practitioner perspectives
Need for Information on Complementary and Alternative Medicine | Day 1
  Interviews between patient and interviewer will help to find out expectations about the need for information on Complementary and Alternative Medicine use from the patient's perspective and from the practitioner's perspective
Improving questionnaire after the practionners' focus group | Day 1
  A practionners' focus group will be organised after the interviews to review the feedbacks and opinions on the questionnaire to improve the questionnaire for the quantitative part of the study

CONTACTS AND LOCATIONS:
Locations (2):
- Reunion (2):
  - CHU La Réunion, Saint-Denis
  - Clinique Saint Clotilde, Sainte-Clotilde

IPD SHARING:
Plan to Share IPD: No